CLINICAL TRIAL: NCT05881070
Title: Effectiveness of Mobile-health Self Management on Quality of Life of Patients Undergoing Chemotherapy
Acronym: MANNER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitas Muhammadiyah Yogyakarta (Other)
Responsible Party: Principal Investigator, Erna Rochmawati, Associate Professor, Universitas Muhammadiyah Yogyakarta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Manner and QOL
Record Dates: First submitted 2023-05-08; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Chemotherapy Effect; Quality of Life; Self Efficacy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile health self-management (Experimental)
  Interventions: Behavioral: Mobile-health self management

INTERVENTIONS:
Behavioral: Mobile-health self management — Mobile-health self management

SUMMARY:
The study will design and evaluate the use of mobile-health based self-management on self-efficacy and quality of life of patients undergoing chemotherapy.

DETAILED DESCRIPTION:
The study will design and evaluate the use of mobile-health based self-management on self-efficacy and quality of life of patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients diagnosed with cancer
* patients who use smart phone

Exclusion Criteria:

* patients with cancer with comorbidity

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient's Quality of life | Four weeks
  The patient's quality of life will be assessed before (T0) and after intervention (T1). The measurement will use EORTC. The score will range from 0-100, where higher score reflects a better quality of life.
Patient's Self-efficacy | four weeks
  The patients self-efficacy will be measured pre and post intervention. The measurement will use the Self-Efficacy for Managing Chronic Disease Scale. The scale has been widely used in cancer setting. Respondents will rate their confidence to perform six self-management behaviours (1 = 'not at all confident' to 10 = 'totally confident'). A mean score is calculated (range 1 to 10). A high score indicates high self-efficacy.

IPD SHARING:
Plan to Share IPD: Undecided